CLINICAL TRIAL: NCT03352024
Title: Impact of Hypno-analgesia, Non-drugs Technique of Care, on Pain That May Inverve During a Lumbar Puncture for Diagnosis of Patient With Mild to Moderate Alzheimer's Dementia.
Brief Title: Impact of Hypno-analgesia on Pain During a Lumbar Puncture for Diagnosis of Alzheimer's Disease
Acronym: PLHYMANEDE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: internal organizational problem and dysfunction of study material
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 9731
Record Dates: First submitted 2017-11-16; First posted 2017-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2017-11

CONDITIONS: Cognitive Impairment; Alzheimer Disease
Keywords: neuro degenerative diseases; Alzheimer's disease; lumbar puncture; CSF; hypno analgesia; no drug care; pain; anxiety; counseling
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Other): Relational care used to help the patient by reducing the fear and anxiety
  Interventions: Other: Relational care
- Hypnosis (Other): Hypno-analgesia is used to help the patient by reducing the fear and anxiety
  Interventions: Other: Hypno-analgesia

INTERVENTIONS:
Other: Relational care — Relational care is combined with a cutaneous anesthesia (Transcutaneous device(plan) of lidocaïne-pilocaïne (EMLA®))
  Arms: Standard Care
Other: Hypno-analgesia — Hypno-analgesia is combined with a cutaneous anesthesia (Transcutaneous device(plan) of lidocaïne-pilocaïne (EMLA®))
  Arms: Hypnosis

SUMMARY:
One of the missions of the Memory of Resources and Research Center (CMRR) is to establish a diagnosis of expertise in patients with amestic, language or behavioral cognitive complaint. Thanks to the dosage of specific biomarkers in the cererbrospinal fluid (CSF), it is currently possible to determine the underlying process of the disease in vivo by assess the pathological amyloid and Tau profile. To obtain these very sensitive and specific biomarkers, clinicians need to perform lumbar puncture (LP). . This exam is easy and reproducible but the gesture image remained negative despite some advances in the materials and care..

Within the Department of Neurology of Montpellier, the recommendations of the Haute Autorité de Santé (HAS) about pain management in adults are applied. A transdermal device of lidocaine-pilocaine (type EMLA) is applied 120 minutes before the LP . In addition, an equimolar oxygen-nitrous oxide (MEOPA) mixture could be added. Then, patients benefit from a helping relationship before and during the gesture dedicated to reduce anxiety.

Until recently, non-medicinal techniques (relaxation, hypnosis ...) were not recommendedin cases of major anxiety or analgesia deemed insufficient. Many studies have shown the efficiency of hypnoalgia in invasive gestures in young children. The University Hospital of Montpellier have developed training about hypnoanalgesia and have been implemented for patients with neurological disorders in our unit. A reduction and even a suppression of pain and a limitation of the apprehension of the gesture have been judged satisfactory both for the patient, the practionner and the nurse practicing regularly the LP. However, this evalusation remained subjective and clinically-based. Thus, it seems relevantto analyse the effect of this technic in order th test the following hypothesis: hypno-analgesia (non-medicinal technique of care) associated with EMLA patch is more effective than the helping relationship associated with EMLA patch to reduce the pain that may inverse during the LP for diagnosis in patient with mild to moderate stage of Alzheimer's disease.

DETAILED DESCRIPTION:
The main objective was to assess whether the use of hypnoanalgesia technic during the LP procedure comparing to commun procedure reduce the pain of the patient evaluated by the hetero-evaluation ALGOPLUS scale.

Secondary objectives were to evaluate the differences between the hypno-analgesia and the helping relationship on:

* pain assessed by the Simple Verbal Scale (EVS);
* pain assessed by the Visual Analog Scale (EVA);
* pain and stress measured by conductance analysis;
* the anxiety score assessed by a STAI self-assessment questionnaire (State-Trait Anxiety Inventory, STAI-Y);
* the rate of failure during the LP procedure.

Methodology :

A monocentric randomized controlled, open-label (with an evaluation of the blind randomization of the randomization arm) with two parallel arms:

* the arm named "hypno-analgesia + EMLA patch" = cutaneous anesthesia associated with hypno-analgesia.
* the arm called "helping relationship + EMLA patch" = cutaneous anesthesia associated with a helping relationship The estimated number of patients was 100. Analysis of the primary outcome measure: The score of the ALGOPLUS scale will compared between the two groups of patients using the Chi2 test after checking the validity conditions of the test.

The project will last 36 months and the duration of the inclusions 24 months. The LP will be carried out during one day of hospitalization as part of the diagnosis assessments. No specific follow-up is scheduled.

ELIGIBILITY:
Inclusion criteria:

* Patient presenting clinical symptoms that may reflect Alzheimer's disease according to the criteria of NIA 2011, with either an isolated hippocampal episodic deficit or associated with dys-executive, phasic or praxic disorders of memory disorder, of insidious progressive evolution with a documented cognitive decline
* Global cognitive score with Mini Mental State MMS between 22 and 27;
* Age between 50 and 90 years ;
* Written and informed consent for this study signed by the patient

Exclusion criteria:

* Refusal to have a LP procedure in the diagnosis process ;
* Refusal to participate in a session of hypno-analgesia;
* Refusal to be filmed during the LP ;
* Patient having already had a session of hypno-analgesia for other diagnostic assessments;
* Patient that done yoga or quite different technique of relaxation ;
* Socio-educational level not allowing the understanding of the neuropsychological tests;
* Not able to follow the majority of the aspects of the study without accompanying ;
* Refusal to sign the written and informed consent ;
* Patient deprived of freedom by court or administrative order

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-11-13 (Estimated)

PRIMARY OUTCOMES:
Algoplus score of pain during the LP procedure | 1 day
  Evaluation of the pain during the Lumbar Punction procedure using the ALGOPLUS (Scale of behavioral evaluation of the pain on 30 points, 30 points being the worst pain) Scale assessment on the patients of each group

SECONDARY OUTCOMES:
Rate of failure of the Lumbar Ponction | 1 day
  This outcome is defined by the incapacity to perform the Lumbar Punction or by the incapacity to collect 12 ml of CSF (cererbrospinal fluid) therefore is defined by the number of the Lumbar Punction aborted
Evaluation of the anxiety | 1 day
  Assessed by an self-completed questionnaire STAI (State-Trait Anxiety Inventory, STAI-Y-A) done before and after the Lumbar Punction and oriented on the anxiety during the LP
Evaluation of the pain | 1 day
  assessed by the Pain monitorTM . The threshold is fixed in 0.2 pic/seconds over whom it is considered that pain is present
Evaluation of the pain by the patient | 1 day
  assessed by the scales EVA (Visual analog scale)
Evaluation of the pain by the patient | 1 day
  assessed by the scales EVS (Simple Verbal scale)

CONTACTS AND LOCATIONS:
Overall Officials: Audrey GABELLE, MD, PhD, Principal Investigator — CHU de Montpellier